CLINICAL TRIAL: NCT01979393
Title: A Randomized Double-blind Phase II Study Evaluating the Role of Maintenance Therapy With Cabozantinib in High Grade Uterine Sarcoma (HGUtS) After Stabilization or Response to Doxorubicin +/- Ifosfamide Following Surgery or in Metastatic First Line Treatment
Brief Title: IRCI Gynae Sarcomas, High Grade Uterine Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gynecologic Oncology Group (Network); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC-62113-55115; 2013-000762-11 (EudraCT Number); UC1306 (Other: GOG)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Uterine Sarcoma
Keywords: Locally advanced; stage III; stage IV; residual disease after primary surgery; newly diagnosed HGUS; Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib (Experimental): Cabozantinib maintenance 60 mg daily for 2 years or until withdrawal criterion After documented disease progression (according to RECIST 1.1), the treatment will be unblinded. Subjects receiving cabozantinib shall be further treated at the investigator discretion.
  Interventions: Drug: Cabozantinib
- Placebo (Experimental): Placebo daily for 2 years or until withdrawal criterion. After documented disease progression (according to RECIST 1.1), the treatment will be unblinded. Subjects receiving placebo shall be offered the option of receiving cabozantinib up to further progression. This is not mandatory and treatment is at the investigator decision.
  Interventions: Drug: Cabozantinib; Drug: Placebo

INTERVENTIONS:
Drug: Cabozantinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate a drug called Cabozantinib which belongs to a family of drugs that have effects on tumour growth, blood supply, invasion and spread.

Therefore, we want to find out whether taking cabozantinib after treatment with surgery and chemotherapy is effective and safe for patients who responded or had stable disease after their chemotherapy.

All participants will receive 4-6 cycles of standard chemotherapy. Those with stabilization or response to the standard chemotherapy will be split into 2 groups (cabozantinib or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are suitable for treatment with doxorubicin +/- ifosfamide and fall within one of the following patient populations:

  • HGUS, HGESS, HGLMS and HG adenosarcoma
  * FIGO stage II and stage III : if adjuvant chemotherapy is proposed
  * FIGO stage IV: if first line chemotherapy is proposed
* Metastatic: diagnosed with disease relapse after local treatment for primary tumor
* at least 18 years old
* written informed consent
* Central pathological confirmation: Histological evidence of HGUS, HGESS, HGLMS and HG adenosarcoma
* Non-progressive patients (CR, PR, SD) at the end of the first line treatment (standard chemotherapy consisting of 4 to 6 cycles of anthracyclines alone or in combination with ifosfamide)
* WHO/ECOG performance status 0-2
* Adequate organ and bone marrow function within 3 days prior to the first dose of study treatment (Cabozantinib/placebo)
* Clinically normal cardiac function
* Women of child bearing potential must have a negative serum/urine pregnancy test within 3 days prior to the first dose of study treatment
* Adequate birth control measures

Exclusion Criteria:

* low-grade ESS, leiomyosarcoma (low or intermediate), carcinosarcoma, low-grade adenosarcoma, rhabdomyosarcoma (alveolar or embryonal) and soft tissue PNET of uterus/cervix.
* contraindications to cabozantinib
* not able to swallow and retain oral tablets
* planned use of chemotherapy, radiation therapy, radionuclide treatment, small molecule tyrosine kinase inhibitor or hormonal therapy, and any other investigational agent (Cabozantinib/placebo) during the treatment period
* concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
* patient with poorly controlled hypertension defined at baseline as blood pressure >150/90
* patients who have suffered a cerebrovascular accident at any time in the past, patients who have suffered a transient ischemic attack in the past 6 months, patients who have suffered a deep venous thrombosis (DVT) or a pulmonary embolism in the past 6 months
* Gastrointestinal disorders
* patients with radiographic evidence of cavitating pulmonary lesion(s)
* patients with tumor in contact with, invading or encasing any major blood vessels
* patients evidence of tumor invading the GI tract
* evidence of active bleeding or bleeding diathesis
* hemoptysis ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment
* signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
* prior major surgery or trauma within 6 weeks prior to first dose of study drug and any wound, fracture, or ulcer should be completely healed
* concurrent or planned treatment with strong inhibitors or inducers of cytochrome P450 3A4/5

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3.5 years from first patient in
  The primary endpoint is PFS rate at 4 months after randomization to cabozantinib or placebo

SECONDARY OUTCOMES:
Progression free survival | 3.5 years from first patient in
Overall survival | 3.5 years from first patient in
Response rate | 3.5 years from first patient in
Duration of response to cabozantinib | 3.5 years from first patient in
Response rate to anthracycline-based chemotherapy for the patients with measurable disease | 3.5 years from first patient in
Assessment of global health status/QoL scale | 3.5 years from first patient in
  The primary health-related quality of life endpoint that is considered of interest for this study is the global health status/QoL scale
Occurence of Adverse Events | 3.5 years from first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Ray-Coquard, MD, Study Chair — Centre Léon Bérard, Lyon, France; Nicholas Reed, MD, Principal Investigator — NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital , Glasgow, United Kingdom
Locations (14):
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Nantes
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands
- Spain (2):
  - Hospital General Vall D'Hebron, Barcelona
  - Hospital Universitario San Carlos, Madrid
- United Kingdom (7):
  - Cambridge University Hospital NHS - Addenbrookes Hospital, Cambridge
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - Royal Marsden Hospital, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Hanvic B, Ray-Coquard I. Gynecological sarcomas: literature review of 2020. Curr Opin Oncol. 2021 Jul 1;33(4):345-350. doi: 10.1097/CCO.0000000000000753. PMID 34009140
- [Derived] Ray-Coquard I, Hatcher H, Bompas E, Casado A, Westermann A, Isambert N, Casali PG, Pratap S, Stark D, Valverde C, Anand A, Huizing M, Floquet A, Lindner L, Hermes B, Seddon B, Coens C, Jones R, Reed N. A randomized double-blind phase II study evaluating the role of maintenance therapy with cabozantinib in high-grade uterine sarcoma after stabilization or response to doxorubicin +/- ifosfamide following surgery or in metastatic first line treatment (EORTC62113). Int J Gynecol Cancer. 2020 Oct;30(10):1633-1637. doi: 10.1136/ijgc-2020-001519. Epub 2020 Jun 15. PMID 32546554